CLINICAL TRIAL: NCT02604953
Title: 1-Year Prospective Study: SD-tVEP and PERG for Early Detection of Retinal Ganglion Cell Dysfunction in Ocular Hypertension Patients
Brief Title: Comparing SD-tVEP and PERG Tests Between Patients With Glaucoma, Patients With High Eye Pressure and "Normal" Patients
Status: Completed | Type: Observational
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, Anand Mantravadi, Principal Investigator, Wills Eye
Other Study IDs: 13-358
Record Dates: First submitted 2015-11-10; First posted 2015-11-16 (Estimated); Last update posted 2017-12-02 (Actual); Status verified 2017-11

CONDITIONS: Glaucoma
Keywords: glaucoma; VEP; PERG; SD-tVEP; ss-PERG
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Ocular Hypertension patients: Ocular hypertension patients are recruited from the Wills Eye Hospital Glaucoma Service. Short Duration Transient Visual Evoked Potential (SD- tVEP) and Pattern electroretinogram (PERG) testing will be conducted.
  Interventions: Diagnostic Test: Short Duration Transient Visual Evoked Potential (SDtVEP); Diagnostic Test: Pattern electroretinogram (PERG)
- Healthy Controls: Healthy adults are recruited from staff, family and friends of Wills Eye Hospital Glaucoma Research Center. Short Duration Transient Visual Evoked Potential (SD- tVEP) and Pattern electroretinogram (PERG) testing will be conducted.
  Interventions: Diagnostic Test: Short Duration Transient Visual Evoked Potential (SDtVEP); Diagnostic Test: Pattern electroretinogram (PERG)
- Glaucoma patients: Glaucoma patients are recruited from the Wills Eye Hospital Glaucoma Service. Short Duration Transient Visual Evoked Potential (SD- tVEP) and Pattern electroretinogram (PERG) testing will be conducted.
  Interventions: Diagnostic Test: Short Duration Transient Visual Evoked Potential (SDtVEP); Diagnostic Test: Pattern electroretinogram (PERG)

INTERVENTIONS:
Diagnostic Test: Short Duration Transient Visual Evoked Potential (SDtVEP) — Short duration transient visual evoked potentials (VEPs) detect disruption of electrical signals at any point along the visual pathway, from the retinal ganglion cells (RGCs) to the primary visual cortex. As an objective measure of visual function, VEP may have advantage over traditional visual field tests, by reducing confounded factors such as age, fatigue, and mental status.
  Other Names: SDtVEP
Diagnostic Test: Pattern electroretinogram (PERG) — Pattern electroretinogram (PERG), an objective test, is used for evaluating early damage to retinal ganglion cells (RGC). In PERG, retinal response is recorded while patterns are viewed in the visual field on a computer monitor.
  Other Names: PERG

SUMMARY:
Wills Eye Hospital Glaucoma Research Center will conduct a 1-year prospective study to assess the ability of a Short Duration Transient Visual Evoked Potential (SD- tVEP) and a Steady-State Pattern electro-retinogram (PERG) vision testing system to detect visual dysfunction in patients with ocular hypertension. The study aims to assess the reversibility of retinal ganglion cell (RGC) dysfunction after administering intraocular pressure (IOP) lowering treatment. The investigators hypothesize that SD-tVEP and PERG testing will help develop better treatment for glaucoma patients by increasing understanding of the physiological relationship of IOP and RGC in glaucomatous injury.

DETAILED DESCRIPTION:
Glaucoma is the most common cause of irreversible blindness worldwide. It is characterized by the progressive loss of retinal ganglion cells (RGCs) and a corresponding loss of vision. Elevated intraocular pressure (IOP) is an important risk factor for glaucoma, but its role in the diagnosis of glaucoma is unclear. Although IOP-lowering therapy delays the onset of glaucoma in some patients with ocular hypertension, even without therapy, 90% of patients will not develop glaucoma over a 5-year period.

Visual evoked potentials (VEPs) are able to detect the disruption of electrical signals at any point along the visual pathway, from the RGCs to the primary visual cortex. As an objective measure of visual function, the VEP may have an advantage over traditional visual field tests, by reducing confounded factors such as age, fatigue, and mental status.

There is a growing body of evidence that SD-tVEP can objectively identify early visual dysfunction due to glaucoma.

Aim 1: Compare the results of the baseline SD-tVEP and PERG vision testing in patients with ocular hypertension to a cohort of 30 healthy subjects and a cohort of 30 patients with glaucoma (of varying severity) to determine its ability to detect visual dysfunction in ocular hypertensive subjects.

Aim 2: Conduct SD-tVEP and PERG testing system in 30 patients with ocular hypertension before and after IOP reduction with topical medication and compare the results of the SD-tVEP and PERG before and after treatment in each patient, to determine its ability to detect reversible RGC dysfunction.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for ocular hypertension patients (Group A):

* Patients diagnosed with ocular hypertension as per the ICD-9 code for ocular hypertension (365.04)
* Age between 21 - 80 years
* IOP more than 21 mm hg in both the eyes.
* Open angles on Gonioscopy
* At least 2 normal and reliable visual fields (Humphrey MD >-2 or Octopus MD ≤0.8; fixation losses, false-positive rate, and false-negative rate each < 33%)
* Normal optic disks, without any of the following signs: rim notches, peripapillary splinter hemorrhages, or C/D asymmetry >0.2 between the two eyes
* BCVA ≥ 20/40, Clear media, Pupil diameter > 3 mm and symmetric
* Spherical refraction within + 5.0 D and cylinder correction within + 3.0 D.

Inclusion Criteria for glaucoma patients (Group B):

* Patients diagnosed with mild, moderate or severe open angle glaucoma as per the (365.xx)
* Age between 21 - 80 years.
* Patients who attend regular follow-up.

Inclusion Criteria for normal subjects (Group C):

* Individuals with no ocular hypertension or any type of glaucoma.
* Available to participate in the study during the required time frame.
* Age 21-80 years.

Exclusion Criteria:

* Incisional eye surgery within the past three months.
* Neurological or musculoskeletal problems that would influence performance on activities of daily living.
* Laser therapy within the previous month.
* Any cause for visual reduction (greater than 20/40 VA) other than glaucoma.
* Any medical condition which in the investigator's opinion would preclude the subject from providing reliable and valid data.
* History of hypersensitivity to Bimatoprost and Brimonidine, or currently taking an MAO inhibitor
* Currently taking any IOP lowering therapies.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Ocular hypertension, glaucoma patients and healthy controls with no eye diseases.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2014-07; Primary Completion 2015-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Short Duration Transient Visual Evoked Potential (SD- tVEP) | 1 day
  Short Duration Transient Visual Evoked Potential (VEP) to objectively measure the functional responses of the entire visual pathway from the anterior segment of the eye to the visual cortex.

CONTACTS AND LOCATIONS:
Overall Officials: Anand Mantravadi, MD, Principal Investigator — Wills Eye Hospital

IPD SHARING:
Plan to Share IPD: No
Data has been presented at the American Glaucoma Society in March 2015 and manuscript will be submitted for publication in 2017.